CLINICAL TRIAL: NCT06022913
Title: Adjunctive Behavioural Activation for Bipolar Depression: A Case Series (BA-BD)
Brief Title: Behavioural Activation for Bipolar Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reykjavik University (Other)
Collaborators: Landspitali University Hospital (Other)
Responsible Party: Principal Investigator, Brynja Bjork Magnusdottir, Assistant professor, Psychologist, Reykjavik University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD0323
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Bipolar Depression
Keywords: Bipolar depression; Bipolar Disorder; Behavioural Activation; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: This is a case series using a multiple baseline design whereby participants are randomly allocated to one of 6 durations of wait at baseline before commencing treatment.
Masking Description: It is not possible to blind the assessor to phase or baseline duration of participants in the case-series, as the length of time between assessments will reveal this. Nevertheless, the assessor and clients will be asked not to disclose which therapist is treating them. Use of self-report measures as the primary outcome measure is intended to minimize potential biases on the side of the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 2 week wait (Other): Participant waits for 2 weeks after their baseline assessment before commencing therapy.
  Interventions: Behavioral: Behavioural Activation (BA)
- 3 week wait (Other): Participant waits for 3 weeks after their baseline assessment before commencing therapy.
  Interventions: Behavioral: Behavioural Activation (BA)
- 4 week wait (Other): Participant waits for 4 weeks after their baseline assessment before commencing therapy.
  Interventions: Behavioral: Behavioural Activation (BA)
- 5 week wait (Other): Participant waits for 5 weeks after their baseline assessment before commencing therapy.
  Interventions: Behavioral: Behavioural Activation (BA)

INTERVENTIONS:
Behavioral: Behavioural Activation (BA) — BA is based on the assumption that depression may be precipitated and is maintained by a reduction in "healthy", adaptive behaviours and positive reinforcement of these, and an increase in avoidance behaviours. Together, these changes reduce the person's immediate distress, often at the expense of their medium and longer term goals. The therapy involves helping the individual to re-establish healthy patterns of activity, and replace avoidance behaviours with more adaptive behaviours that are constructive in the longer term.
  The intervention consists of up to 20 individual therapy sessions of Behavioural Activation, with one booster session three months after the end of therapy. Each session lasts approximately 50 minutes and this is supplemented by home practice between sessions.

SUMMARY:
Bipolar disorder (BD) affects between 1-3% of the world's population. People with BD experience episodes of mania or hypomania and in most cases, they experience periods of depression which can cause difficulties in daily life. Psychological therapies for people experiencing depression without mania or hypomania are widely available, but there is little research into how effective these therapies are for people with BD. Behavioral activation therapy (BA) is based on behavioral theory and has been proven to be an effective treatment for unipolar depression. It helps people re-establish healthier activity patterns and sleep regulation, especially in BD for mood stabilization. BA is theoretically and clinically well matched to the treatment of bipolar depression, but there is still very little research into offering BA to people with BD.

The first aim of the current research is to implement BA for people with depression in Bipolar Disorder and study if it is feasible for this patient group. The second aim is to do a pilot study on the effectiveness of the treatment for this patient group. The research will be implemented with people seeking treatment at the specialized service for bipolar disorder at Landspítali University Hospital in Iceland. The participants will receive treatment as usual and the BA will be adjunctive.

At least ten people, that are currently experiencing Bipolar Depression and are willing to take part, will receive up to 20 individual therapy sessions of BA that have been adapted for Bipolar Depression (BA-BD), and will complete regular questionnaires and interviews.

The study will be a replication study to validate the previous study's findings by Kim, W. et al., 2022 in another setting.

ELIGIBILITY:
Inclusion Criteria:

* scoring in the clinical range on a self-report measure of depression severity (the PHQ-9) meeting diagnostic criteria for depression based on a diagnosis on Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND)

meeting diagnostic criteria for Bipolar I or II Disorder DIAMOND) participants will require a working knowledge of written and spoken Icelandic, sufficient to make use of therapy and complete research assessments without the need for a translator.

Exclusion Criteria:

* current/past learning disability, organic brain change, substance dependence (drugs and alcohol) that would compromise the ability to use therapy
* current marked risk to self (i.e., self-harm or suicide) that we deem could not be appropriately managed in the Bipolar outpatient clinic at Landspitali.
* currently lacking the capacity to give informed consent
* currently receiving other psychosocial therapy for depression or bipolar disorder
* presence of another area of difficulty that the therapist and client believe should be the primary focus of intervention (for example, Post-Traumatic Stress Disorder, psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimally clinically significant improvement in depression symptoms for a majority of participants (>60%) | through study completion, an average of 7 months
  Participants' weekly completion of the Patient Health Questionnaire-9 (PHQ-9)
Therapy uptake rate | through study completion, an average of 7 months
  Number of participants randomised who attend at least 1 treatment session
Therapy completion rate | through study completion, an average of 7 months
  Proportion of participants that attend at least 8 treatment sessions
Change in activity levels as measured by consumer connected health devices | through study completion, an average of 7 months
  Measures of activity levels as by Withings health devices
Change in Sleep Duration measured by health device | through study completion, an average of 7 months
  Measures of sleep duration by Withings health devices
No significant adverse reaction for participants | through study completion, an average of 7 months
  Participant reports of adverse events elicited by researchers and therapists

SECONDARY OUTCOMES:
Altman Self-Rating Mania Scale (ASRM) | 1 week
  5 item self-report measure of hypomania symptoms over the past week
Work and Social Adjustment Scale (WSAS) | 24 hours
  5 item self-report scale of functional impairment attributable to an identified problem
Hamilton Depression Scale (HAM-D) | 1 week
  17 item observer-rated scale measuring symptoms of depression over the past week
Brief Quality of Life in Bipolar Disorder (Brief QoLBD) | 1 week
  12 item self-report measure of disorder-specific quality of life
General Anxiety Disorder Assessment - 7 (GAD7) | 2 weeks
  7 item self-report measure of anxiety symptoms
Behavioral Activation for Depression Scale (BADS) | 1 week
  25 item self-report measure of changes in activation and avoidance over the past week
Snaith-Hamilton Pleasure Scale (SHAPS) | 1 week
  14 item self-report measure of level of anhedonia
Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND) | Six months
  Standardized interview to establish whether the participant meets research diagnostic criteria for lifetime Bipolar I or II Disorder, current depressive episode, and to establish whether they are experiencing current substance dependence
Young mania rating scale | 48 hours
  11 item observer-rated scale measuring the severity of manic states
Six daily questions | 24 hours
  Six daily questions in mobile about goal achievement, mood, sleep etc
The Quality of Behavioral Activation Scale (Q-BAS) | 1 week
  To assess the quality of and adherence to BA clinical protocol using audiotapes of therapy sessions

CONTACTS AND LOCATIONS:
Overall Officials: Brynja B Magnúsdóttir, PhD, Study Chair — Reykjavik University; Anna S Islind, PhD, Principal Investigator — Reykjavik University; Steinunn G Sigurðardóttir, MSc, Principal Investigator — Reykjavik University
Locations (1):
- Landspitali university hospital, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: Yes
All data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Access will be possible from the date of publication.
Access Criteria: The dataset will be anonymous and registered with a metadata-only record, allowing the research team to control access to the dataset, and restricting it to appropriately qualified third parties.